CLINICAL TRIAL: NCT01478971
Title: A Phase 3b Single-Arm, Conversion Study From Epoetin Alfa to Monthly Peginesatide Injection in Patients With Chronic Kidney Disease on Dialysis
Brief Title: Conversion Study From Epoetin Alfa to Monthly Peginesatide Injection in Patients With Chronic Kidney Disease on Dialysis
Acronym: DIAMOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-18; U1111-1150-2575 (Registry Identifier: WHO)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Anemia; Chronic Renal Failure; CRF; Chronic Kidney Disease; CKD; Erythropoietin; Hematide; Peginesatide; Hemoglobin; Hgb; Red Blood Cell; Red Blood Cell Production; Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia; Kidney Failure, Chronic | interventions — Erythropoietin; peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- peginesatide injection (Experimental): In the first 6 months participants received standard of care treatment with epoetin (the Standard of Care Period [SCP]), followed by a 1-week erythropoiesis-stimulating agent (ESA)-Free Period, followed by peginesatide injection for 6 months (the Peginesatide Treatment Period [PTP]).
  Interventions: Drug: Epoetin; Drug: Peginesatide

INTERVENTIONS:
Drug: Epoetin — Commercially available epoetin alfa administered weekly, twice weekly, or thrice weekly at an initial starting dose, frequency of administration, and mode of administration (intravenous [IV] or subcutaneous [SC]) individually determined for each participant using the site's usual standard of care. Subsequent dose adjustments or dose holds may have been made in order to maintain a hemoglobin concentration of <11 g/dL.
Drug: Peginesatide — Administered as a once monthly intravenous (IV) or subcutaneous (SC) injection. The initial dose of peginesatide injection was based on the final weekly dose of epoetin administered in the SCP; subsequent doses may have been adjusted in order to maintain hemoglobin concentrations at <11 g/dL.
  Other Names: Omontys

SUMMARY:
The purpose of this study is to understand the effects of a dialysis center switching its dialysis patients from using Epoetin alfa to peginesatide injection on hemoglobin levels and other parameters.

DETAILED DESCRIPTION:
Monthly Erythropoiesis-Stimulating Agents (ESA) dosing, compared with the longstanding practice of dosing three times per week, represents a significant change in anemia treatment for dialysis patients. Because of the differences in the processes needed to support monthly dosing versus thrice weekly dosing, there is a need to prospectively identify and evaluate factors in the dialysis environment during center-level transition of patients from one ESA to another.

AFX01-18 is a Phase 3b open-label, single-arm conversion study that was conducted at 5 hemodialysis sites in the United States, and enrolled Chronic Kidney Disease (CKD) patients receiving outpatient, in-center hemodialysis. The study treatment period was approximately 12 months in duration. Participants received peginesatide injection for approximately six months.

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent in accordance with institutional, local, and national guidelines
* Are ≥18 years of age at the start of screening
* Have been on in-center hemodialysis for ≥12 weeks at the start of screening
* Are currently maintained on Epoetin at the start of screening
* If sexually active and a female of childbearing potential, are willing to use highly effective method of birth control ≥4 weeks before study enrollment and through the study
* If a female of childbearing potential, have a negative pregnancy test during screening

Exclusion Criteria:

* Are scheduled for a renal transplantation during study (Note: patients awaiting transplantation with no date scheduled may enroll.)
* Have an active malignancy or malignancy treated within one year prior to the start of screening for curative or palliative intent (Note: patients with non-melanoma skin cancers may enroll.)
* Have known intolerance to any ESA or PEGylated molecule
* Have been exposed to any investigational agent during the four weeks prior to the start of screening or are anticipated to receive such agents during the study
* Have any significant medical or psychiatric condition judged by the investigator to prevent informed consent or study compliance
* Are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (5):
- United States (5):
  - Research Facility, Sacramento, California
  - Research Facility, San Diego, California
  - Research Facility, San Jose, California
  - Research Facility, North Brunswick, New Jersey
  - Research Facility, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 11 October 2011 to 08 February 2013.
Pre-assignment Details: Participants with chronic kidney disease and on dialysis continued to receive their standard of care epoetin treatment for 6 months and then transitioned to receive peginesatide injection for 6 months.
Groups:
- Peginesatide Injection: In the first 6 months participants received Standard of Care treatment with epoetin (the Standard of Care Period [SCP]), followed by a 1 -week erythropoiesis-stimulating agent (ESA)-free period, followed by a transition to once monthly peginesatide injection for 6 months (the Peginesatide Treatment Period [PTP]).
Period: Standard of Care Period
Arm/Group | Peginesatide Injection
Started | 184
Received Treatment | 178
Completed | 159
Not Completed | 25
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Death | 8
Not completed — Lost to Follow-up | 9
Not completed — Other | 4
Period: Peginesatide Treatment Period
Arm/Group | Peginesatide Injection
Started | 157 (2 participants terminated the study before transitioning to peginesatide for unknown reasons)
Completed | 143
Not Completed | 14
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 4
Not completed — Lost to Follow-up | 4
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Arm/Group | Peginesatide Injection
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (15.33)
Age, Customized [Number; unit: participants]
  < 65 years | 103
  65 - 74 years | 44
  ≥ 75 years | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 94
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 76
  Not Hispanic or Latino | 102
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Black | 43
  Native Hawaiian or Other Pacific Islander | 5
  White | 119
Region of Enrollment [Number; unit: participants]
  United States | 178 (3.71)
Weight [Mean (Standard Deviation); unit: kg] — Weight data only available for 177 participants.
  kg | 83.8 (22.93)
Time on dialysis [Mean (Standard Deviation); unit: years] | 4.2 (3.71)
Kidney transplant recipient [Number; unit: participants]
  Yes | 17
  No | 161
Nephrotic syndrome history [Number; unit: participants]
  Yes | 30
  No | 148
Primary cause of chronic kidney disease [Number; unit: participants]
  Diabetes | 97
  Hypertension | 37
  Cystic renal disease | 6
  Interstitial nephritis | 2
  Glomerulonephritis | 15
  Urological | 4
  Immunoglobulin (Ig) A nephropathy | 3
  Congenital | 1
  Unknown | 3
  Other | 10
Current dialysis frequency [Number; unit: participants]
  2 times a week | 3
  3 times a week | 169
  4 times a week | 4
  5 times a week | 1
  6 times a week | 1
Baseline hemoglobin [Mean (Standard Deviation); unit: g/dL] | 10.9 (0.96)
Ferritin [Mean (Standard Deviation); unit: ng/mL] — Ferritin data only available for 149 participants.
  ng/mL | 1068.7 (513.1)
Transferrin saturation [Mean (Standard Deviation); unit: percent saturation] — Transferrin saturation data only available for 146 participants.
  percent saturation | 35.2 (13.85)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Undergoing Conversion to Peginesatide Injection
Time Frame: 6 months
Population: All participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide Injection
Number analyzed (Participants) | 178
percentage of participants | 88

2. Secondary Outcome: Peginesatide Dosing
Description: The starting dose, mean dose throughout the study, and mean dose during the last week of treatment of peginesatide.
Time Frame: Month 6 - 12
Population: Participants who received at least 1 dose of study treatment during the Peginesatide Treatment Period.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Peginesatide Injection
Number analyzed (Participants) | 157
mg
  Starting Dose | 5.1 (2.82)
  Average Dose During Treatment Period | 4.9 (2.97)
  Last Weekly Average Dose | 5.2 (3.68)

3. Secondary Outcome: Peginesatide Dose Deviations
Description: Data collected by sponsor of study (Affymax), and sponsor did not provide aggregate summary data.
Time Frame: Months 6 - 12
Arm/Group | Peginesatide Injection
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Hemoglobin Levels Greater Than 10 and Less Than or Equal to 11 g/dL
Description: Percentage of participants with hemoglobin values within the hemoglobin range of 10-11 g/dL.
Time Frame: Months 1, 2, 3, 4, 5 and 6 of each treatment period
Population: Full Analysis Population included all enrolled participants who received at least 1 dose of study treatment during the Peginesatide Treatment Period. n indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Groups:
- Epoetin Standard of Care: In the first 6 months participants received Standard of Care treatment with epoetin (the Standard of Care Period [SCP]).
- Peginesatide Treatment Period: In the second six months of the study participants transitioned to peginesatide injection (the Peginesatide Treatment Period [PTP]).
Arm/Group | Epoetin Standard of Care | Peginesatide Treatment Period
Number analyzed (Participants) | 157 | 157
percentage of participants
  Month 1 (n=156, 155) | 39.1 | 44.5
  Month 2 (n=157, 155) | 40.8 | 46.5
  Month 3 (n=156, 155) | 41.0 | 45.2
  Month 4 (n=156, 151) | 44.9 | 49.0
  Month 5 (n=157, 147) | 42.7 | 44.9
  Month6 (n=157, 146) | 58.0 | 39.0

5. Secondary Outcome: Percentage of Participants Who Received at Least One Intravenous Iron Dose
Description: Participants received iron supplementation during the study to prevent iron deficiency and to maintain iron stores.
Time Frame: 12 months
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Standard of Care | Peginesatide Treatment Period
Number analyzed (Participants) | 178 | 157
percentage of participants | 85.4 | 73.2

6. Secondary Outcome: Percentage of Participants Who Received a Whole Blood or Red Blood Cell Transfusion
Time Frame: 12 months
Population: Safety population
Measure: Number; unit: percentage of participants
Arm/Group | Epoetin Standard of Care | Peginesatide Treatment Period
Number analyzed (Participants) | 178 | 157
percentage of participants | 10.7 | 8.3

ADVERSE EVENTS:
Time Frame: 12 months plus 4 to 5 weeks after the last dose of study treatment or last visit.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- ESA Free Week: A one-week erythropoiesis-stimulating agent (ESA)-free period following 6 months of standard of care.
- Peginesatide Treatment Period: In the second six months of the study participants transitioned to once monthly peginesatide injection (the Peginesatide Treatment Period [PTP]).
Arm/Group | Epoetin Standard of Care | ESA Free Week | Peginesatide Treatment Period
Serious Adverse Events (participants affected / at risk) | 64/178 | 2/160 | 54/157
Other Adverse Events (participants affected / at risk) | 74/178 | 7/160 | 70/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Standard of Care (N=178) | ESA Free Week (N=160) | Peginesatide Treatment Period (N=157)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 5 | 0 | 6
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 4
Acute myocardial infarction (Cardiac disorders) | 4 | 0 | 2
Cardiac arrest (Cardiac disorders) | 3 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 2
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 3
Ascites (Gastrointestinal disorders) | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 5 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 1
Device malfunction (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 0 | 2
Sepsis (Infections and infestations) | 6 | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 0 | 0
Gangrene (Infections and infestations) | 3 | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 1 | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 2
Cellulitis (Infections and infestations) | 2 | 1 | 1
Device related sepsis (Infections and infestations) | 2 | 0 | 0
Infectious peritonitis (Infections and infestations) | 2 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cholangitis suppurative (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1 | 5
Fluid overload (Metabolism and nutrition disorders) | 4 | 1 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 3 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 4
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 3 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 4
Hypotension (Vascular disorders) | 2 | 0 | 3
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Diabetic foot (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Gallbladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 2
Brachiocephalic vein stenosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Standard of Care (N=178) | ESA Free Week (N=160) | Peginesatide Treatment Period (N=157)
Anaemia (Blood and lymphatic system disorders) | 13 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 12 | 1 | 12
Vomiting (Gastrointestinal disorders) | 10 | 2 | 9
Abdominal pain upper (Gastrointestinal disorders) | 9 | 0 | 3
Nausea (Gastrointestinal disorders) | 9 | 1 | 6
Nasopharyngitis (Infections and infestations) | 9 | 1 | 4
Fall (Injury, poisoning and procedural complications) | 10 | 0 | 16
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 15 | 2 | 10
Hyperphosphataemia (Metabolism and nutrition disorders) | 7 | 1 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 1 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 0 | 7
Headache (Nervous system disorders) | 7 | 1 | 13
Dizziness (Nervous system disorders) | 7 | 0 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.